CLINICAL TRIAL: NCT02389452
Title: A Multicenter, Prospective, Open-Label Study of the Safety and Efficacy of 6 mL Synvisc-One ® (Hylan G F 20) in Indian Patients With Symptomatic Osteoarthritis of the Knee(s) After Initial and Repeat Treatment
Brief Title: Study of Safety and Efficacy of 6 mL Synvisc-One (Hylan G-F 20) in Indian Patients With Symptomatic Osteoarthritis of Knee(s) After Initial and Repeat Treatment
Acronym: OASIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYNV03809; U1111-1167-6813 (Other: World Health Organization)
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — hylan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Synvisc-One (Experimental): Single 6 mL IA injection of Synvisc-One (48 mg of cross-linked hylan polymer) at Day 0 (Initial Treatment). Participants received repeat injection based on physician's discretion of safety and efficacy (no major safety concerns and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) A1 subscore [measurement of pain while walking on flat surface] between 40-80 mm, measured on a 0-100 mm scale with 0 represents no pain and 100 represents worst possible pain) at Week 26, 39 or 52 (Repeat treatment).
  Interventions: Drug: Synvisc-One

INTERVENTIONS:
Drug: Synvisc-One — intraarticular injection
  Other Names: GZ402662; hylan G-F 20

SUMMARY:
Primary Objective:

To evaluate the safety and efficacy of a single 6 mL intraarticular (IA) injection of Synvisc-One in participants in India with symptomatic osteoarthritis (OA) of the knee(s).

Secondary Objective:

To evaluate the safety and short-term efficacy of a repeat treatment with Synvisc-One.

DETAILED DESCRIPTION:
A period of approximately 19 months was anticipated from the time the first participants was enrolled in the study to the completion of the study (last participant out). Individual participant participation lasted from 7 to 13 months depending on the timing of repeat treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participant aged 30 years or older, with active lifestyle.
* The participant must be able to read, understand, and sign an informed consent form, understand requirements for followup visits, and must be willing to provide information at the scheduled evaluations.
* The participant had a diagnosis of OA of the target knee confirmed by recent X-ray (mild to moderate joint space narrowing and/or osteophytes (ie, Kellgren Lawrence [KL] Grade I-III), predominant in the tibiofemoral compartment.
* WOMAC A1 baseline 100 mm visual analog scale (VAS) score from 40-80 mm (moderate or severe walking pain) in the target knee.
* Participants with bilateral disease may be included in the study with the below strict conditions:

  * Only one knee included in the efficacy assessment and considered the target knee (the worst knee by the WOMAC A1 pain scale should be selected). The selected knee must meet the inclusion and exclusion criteria.
  * The non-target knee may also be treated with Synvisc-One and does not need to meet the KL grade knee specific inclusion criteria described above. The other criteria do apply.
* If female, must had a negative urine pregnancy test and continue to use a medically acceptable form of contraception for the duration of the study. Otherwise, females must had been surgically sterile or postmenopausal (as documented in the medical history) for at least 1 year.

Exclusion Criteria:

* Significant (requiring surgical correction) valgus or varus deformity of the knee, ligamentous laxity, or meniscal instability.
* Concomitant inflammatory or any other disease/condition which may affect joints (eg, rheumatoid arthritis, metabolic bone disease, psoriasis, gout, pseudogout, or chondrocalcinosis).
* History of sepsis in any joint or any clinical concern for a subacute infectious process in the target joint.
* History of surgery in the target knee.
* Planned surgery on any lower extremity joint.
* Clinically significant venous or lymphatic stasis present in the leg(s).
* Clinically apparent tense effusion or inflammation at the target knee.
* Skin disease or infection in the area of the injection site.
* Any musculoskeletal condition that would impede measurement of efficacy at the target knee.
* Pregnant or lactating women.
* Hypersensitivities to avian proteins and/or any components of hyaluronan-based injection.
* Treatment with any hyaluronic acid (HA) or derivatives in the previous 6 months.
* Treatment with IA steroids in the previous 3 months.
* Any contraindication to IA injection, eg, anticoagulant therapy or clinical concern for potential coagulopathy (eg, liver disease).
* Any significant medical condition (eg, significant psychiatric or neurological disorders or active alcohol/drug abuse), any medical condition that is unstable/poorly controlled or other factors (eg, planned relocation) that the Investigator felt would interfere with study evaluations and study participation.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 36 sites in India between February 16, 2010 and September 7, 2011.
Groups:
- Synvisc-One: Single 6 mL intra-articular (IA) injection of Synvisc-One (48 mg of cross-linked hylan polymer) at Day 0 (Initial Treatment). Participants received repeat injection based on physician's discretion of safety and efficacy at Week 26, 39 or 52 (Repeat treatment). Repeat injection was given if there was no major safety concerns and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) A1 subscore (measurement of pain while walking on flat surface) was between 40-80 mm (at Week 26, 39 or 52 ) when measured on a 0-100 mm scale, where higher score indicate higher pain.
Period: Overall Study
Arm/Group | Synvisc-One
Started | 394
Participants Received Repeat Injection | 11 (Repeat injection based on physician's assessment of efficacy and safety at Week 26, 39 or 52.)
Completed | 369
Not Completed | 25
Not completed — Lost to Follow-up | 13
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 5
Not completed — Enrolled but Not Eligible for Study | 6

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all participants who received at least one dose of study medication.
Groups:
- Synvisc-One: Single 6 mL IA injection of Synvisc-One at Day 0 (Initial Treatment). Participants received repeat injection based on physician's discretion of safety and efficacy at Week 26, 39 or 52 (Repeat treatment). Repeat injection was given if there was no major safety concerns and WOMAC A1 subscore (measurement of pain while walking on flat surface) was between 40-80 mm (at Week 26, 39 or 52) when measured on a 0-100 mm scale, where higher score indicate higher pain.
Arm/Group | Synvisc-One
Number analyzed (Participants) | 394
Age, Continuous [Mean (Standard Deviation); unit: years] — Number of participants analysed for this parameter were 392.
  years | 57.6 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285
  Male | 109
Weight [Mean (Standard Deviation); unit: kilograms] | 70.72 (11.526)
Height [Mean (Standard Deviation); unit: centimeters] | 160.11 (8.836)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] | 27.66 (4.477)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in WOMAC A1 Subscore at Week 26
Description: WOMAC is health status measure questionnaire comprising 3 subscales (pain, stiffness and physical function). WOMAC A1 (measure of pain during walking on a flat surface) was measured using a visual analogue scale (100 mm line marked by participants with total score ranging from 0-100). Lower score represents lower pain.
Time Frame: Baseline, Week 26 (missing data imputed by Last Observation Carried Forward [LOCF]).
Population: ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc-One
Number analyzed (Participants) | 394
units on a scale | -28.0 (19.89)
Statistical Analysis 1: Comparison: Synvisc-One; Test type: Superiority or Other; p < 0.0001, Paired t-test

2. Secondary Outcome: Change From Baseline in WOMAC A1 Subscore at Week 52
Description: as for outcome 1
Time Frame: Baseline, Week 52 (missing data imputed by LOCF)
Population: ITT population. Number of participants analyzed=participants with baseline and Week 52 data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc-One
Number analyzed (Participants) | 388
units on a scale | -32.7 (19.95)

3. Secondary Outcome: Change From Baseline in WOMAC A Score at Week 52
Description: WOMAC is health status measure questionnaire comprising 3 subscales (pain, stiffness and physical function). WOMAC A (measure of pain) calculated as a mean of 5 individual components, measured using a visual analogue scale (100 mm line marked by participants with score ranging from 0-100). Total score range is 0 to 100, where higher scores indicate higher pain.
Time Frame: Baseline, Week 52 (missing data imputed by LOCF)
Population: ITT population. Number of participants analyzed=participants with baseline and Week 52 data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc-One
Number analyzed (Participants) | 388
units on a scale | -29.18 (19.158)

4. Secondary Outcome: Change From Baseline in WOMAC B Score at Week 52
Description: WOMAC is health status measure questionnaire comprising 3 subscales (pain, stiffness and physical function). WOMAC B (measure of stiffness) calculated as a mean of 2 individual components, measured using a visual analogue scale (100 mm line marked by participants with score ranging from 0-100). Total score range is 0 to 100, where higher scores indicate higher stiffness. Stiffness is defined as a sensation of decreased ease in movement of joint.
Time Frame: Baseline, Week 52 (missing data imputed by LOCF)
Population: ITT population. Number of participants analyzed=participants with baseline and Week 52 data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc-One
Number analyzed (Participants) | 388
units on a scale | -25.77 (22.047)

5. Secondary Outcome: Change From Baseline in WOMAC C Score at Week 52
Description: WOMAC is health status measure questionnaire comprising 3 subscales (pain, stiffness and physical function). WOMAC C (measure of physical function) calculated as a mean of 17 individual components, measured using a visual analogue scale (100 mm line marked by participants with score ranging from 0-100). Total score range is 0 to 100, where higher scores indicate higher worse function. Physical function refers to participant's ability to move around and perform usual activities of daily living.
Time Frame: Baseline, Week 52 (missing data imputed by LOCF)
Population: ITT population. Number of participants analyzed=participants with baseline and Week 52 data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc-One
Number analyzed (Participants) | 388
units on a scale | -25.72 (19.449)

6. Secondary Outcome: Patient Global Assessment (PTGA) Score at Week 52
Description: PTGA (global self-assessment of target knee osteoarthritis condition) was measured using the 5 point Likert scale (0=very well, 1=well, 2=fair, 3=poor, 4=very poor) by participants to rate the osteoarthritis condition. Number of participants with different categories of PTGA score at Week 52 are reported.
Time Frame: Week 52 (missing data imputed by LOCF)
Population: ITT population. Number of participants analyzed=participants with baseline and Week 52 data.
Measure: Number; unit: participants
Arm/Group | Synvisc-One
Number analyzed (Participants) | 388
participants
  Very well | 82
  Well | 175
  Fair | 90
  Poor | 40
  Very poor | 1

7. Secondary Outcome: Clinician Observer Global Assessment (COGA) Score at Week 52
Description: COGA (global self-assessment of target knee osteoarthritis condition) was measured using the 5 point Likert scale (0=very well, 1=well, 2=fair, 3=poor, 4=very poor) by the physician to rate participant's osteoarthritis condition. Number of participants with different categories of PTGA score at Week 52 are reported.
Time Frame: Week 52 (missing data imputed by LOCF).
Population: ITT population. Number of participants analyzed=participants with baseline and Week 52 data.
Measure: Number; unit: participants
Arm/Group | Synvisc-One
Number analyzed (Participants) | 388
participants
  Very well | 77
  Well | 177
  Fair | 98
  Poor | 35
  Very poor | 1

8. Secondary Outcome: 12-Item Short Form Health Survey (SF-12)
Description: SF-12 health survey is a self-reported questionnaire to measure participant's profile of functional health and well-being. It includes following 12 questions (Q): Q1 In general, health status; Q2a Limitation of moderate activities; Q2b Limitation of climbing; Q3a Less accomplishment due to physical health; Q3b Limited in the kind of work or other activities due to physical health; Q4a Less accomplishment due to emotional problems; Q4b Did work or other activities less carefully than usual due to emotional problems; Q5 Pain interfere with normal work; Q6a Felt calm and peaceful; Q6b Had lot of energy; Q6c Felt downhearted and low; and Q7 Physical health or emotional problems interfered with social activities. Number of participants with response to each Q are reported.
Time Frame: Baseline, Week 26, 52
Population: ITT population. Number of participants evaluable for baseline, Week 26 and Week 52 were 394, 394 and 388, respectively.
Measure: Number; unit: participants
Arm/Group | Synvisc-One
Number analyzed (Participants) | 394
participants
  Q1: Excellent/Very Good, Baseline | 35
  Q1: Excellent/Very Good, Week 26 | 87
  Q1: Excellent/Very Good, Week 52 | 135
  Q1: Good, Baseline | 139
  Q1: Good, Week 26 | 230
  Q1: Good, Week 52 | 189
  Q1: Fair/Poor, Baseline | 219
  Q1: Fair/Poor, Week 26 | 76
  Q1: Fair/Poor, Week 52 | 64
  Q1: Missing, Baseline | 1
  Q1: Missing, Week 26 | 1
  Q1: Missing, Week 52 | 0
  Q2a: Yes, Limited a Lot/a Little, Baseline | 367
  Q2a: Yes, Limited a Lot/a Little, Week 26 | 303
  Q2a: Yes, Limited a Lot/a Little, Week 52 | 293
  Q2a: No Not Limited at All, Baseline | 24
  Q2a: No Not Limited at All, Week 26 | 90
  Q2a: No Not Limited at All, Week 52 | 95
  Q2a: Missing, Baseline | 3
  Q2a: Missing, Week 26 | 1
  Q2a: Missing, Week 52 | 0
  Q2b: Yes, Limited a Lot/a Little, Baseline | 373
  Q2b: Yes, Limited a Lot/a Little, Week 26 | 338
  Q2b: Yes, Limited a Lot/a Little, Week 52 | 334
  Q2b: No Not Limited at All, Baseline | 19
  Q2b: No Not Limited at All, Week 26 | 55
  Q2b: No Not Limited at All, Week 52 | 54
  Q2b: Missing, Baseline | 2
  Q2b: Missing, Week 26 | 1
  Q2b: Missing, Week 52 | 0
  Q3a: All/Most of the Time, Baseline | 152
  Q3a: All/Most of the Time, Week 26 | 62
  Q3a: All/Most of the Time, Week 52 | 76
  Q3a: Some of the Time, Baseline | 163
  Q3a: Some of the Time, Week 26 | 170
  Q3a: Some of the Time, Week 52 | 142
  Q3a: A Little/None of the Time, Baseline | 76
  Q3a: A Little/None of the Time, Week 26 | 159
  Q3a: A Little/None of the Time, Week 52 | 169
  Q3a: Missing, Baseline | 3
  Q3a: Missing, Week 26 | 3
  Q3a: Missing, Week 52 | 1
  Q3b: All/Most of the Time, Baseline | 137
  Q3b: All/Most of the Time, Week 26 | 58
  Q3b: All/Most of the Time, Week 52 | 57
  Q3b: Some of the Time, Baseline | 158
  Q3b: Some of the Time, Week 26 | 147
  Q3b: Some of the Time, Week 52 | 148
  Q3b: A Little/None of the Time, Baseline | 96
  Q3b: A Little/None of the Time, Week 26 | 187
  Q3b: A Little/None of the Time, Week 52 | 183
  Q3b: Missing, Baseline | 3
  Q3b: Missing, Week 26 | 2
  Q3b: Missing, Week 52 | 0
  Q4a: All/Most of the Time, Baseline | 114
  Q4a: All/Most of the Time, Week 26 | 60
  Q4a: All/Most of the Time, Week 52 | 58
  Q4a: Some of the Time, Baseline | 149
  Q4a: Some of the Time, Week 26 | 115
  Q4a: Some of the Time, Week 52 | 132
  Q4a: A Little/None of the Time, Baseline | 128
  Q4a: A Little/None of the Time, Week 26 | 217
  Q4a: A Little/None of the Time, Week 52 | 198
  Q4a: Missing, Baseline | 3
  Q4a: Missing, Week 26 | 2
  Q4a: Missing, Week 52 | 0
  Q4b: All/Most of the Time, Baseline | 88
  Q4b: All/Most of the Time, Week 26 | 48
  Q4b: All/Most of the Time, Week 52 | 56
  Q4b: Some of the Time, Baseline | 166
  Q4b: Some of the Time, Week 26 | 131
  Q4b: Some of the Time, Week 52 | 128
  Q4b: A Little/None of the Time, Baseline | 137
  Q4b: A Little/None of the Time, Week 26 | 213
  Q4b: A Little/None of the Time, Week 52 | 204
  Q4b: Missing, Baseline | 3
  Q4b: Missing, Week 26 | 2
  Q4b: Missing, Week 52 | 0
  Q5: Not at All/A Little Bit, Baseline | 70
  Q5: Not at All/A Little Bit, Week 26 | 207
  Q5: Not at All/A Little Bit, Week 52 | 219
  Q5: Moderately, Baseline | 182
  Q5: Moderately, Week 26 | 122
  Q5: Moderately, Week 52 | 105
  Q5: Quite a Bit/Extremely, Baseline | 140
  Q5: Quite a Bit/Extremely, Week 26 | 63
  Q5: Quite a Bit/Extremely, Week 52 | 64
  Q5: Missing, Baseline | 2
  Q5: Missing, Week 26 | 2
  Q5: Missing, Week 52 | 0
  Q6a: All/Most of the Time, Baseline | 188
  Q6a: All/Most of the Time, Week 26 | 240
  Q6a: All/Most of the Time, Week 52 | 244
  Q6a: Some of the Time, Baseline | 112
  Q6a: Some of the Time, Week 26 | 106
  Q6a: Some of the Time, Week 52 | 121
  Q6a: A Little/None of the Time, Baseline | 92
  Q6a: A Little/None of the Time, Week 26 | 46
  Q6a: A Little/None of the Time, Week 52 | 23
  Q6a: Missing, Baseline | 2
  Q6a: Missing, Week 26 | 2
  Q6a: Missing, Week 52 | 0
  Q6b: All/Most of the Time, Baseline | 122
  Q6b: All/Most of the Time, Week 26 | 190
  Q6b: All/Most of the Time, Week 52 | 215
  Q6b: Some of the Time, Baseline | 154
  Q6b: Some of the Time, Week 26 | 134
  Q6b: Some of the Time, Week 52 | 132
  Q6b: A Little/None of the Time, Baseline | 115
  Q6b: A Little/None of the Time, Week 26 | 67
  Q6b: A Little/None of the Time, Week 52 | 40
  Q6b: Missing, Baseline | 3
  Q6b: Missing, Week 26 | 3
  Q6b: Missing, Week 52 | 1
  Q6c: All/Most of the Time, Baseline | 67
  Q6c: All/Most of the Time, Week 26 | 28
  Q6c: All/Most of the Time, Week 52 | 53
  Q6c: Some of the Time, Baseline | 162
  Q6c: Some of the Time, Week 26 | 102
  Q6c: Some of the Time, Week 52 | 107
  Q6c: A Little/None of the Time, Baseline | 159
  Q6c: A Little/None of the Time, Week 26 | 261
  Q6c: A Little/None of the Time, Week 52 | 227
  Q6c: Missing, Baseline | 6
  Q6c: Missing, Week 26 | 3
  Q6c: Missing, Week 52 | 1
  Q7: All/Most of the Time, Baseline | 116
  Q7: All/Most of the Time, Week 26 | 35
  Q7: All/Most of the Time, Week 52 | 43
  Q7: Some of the Time, Baseline | 166
  Q7: Some of the Time, Week 26 | 129
  Q7: Some of the Time, Week 52 | 119
  Q7: A Little/None of the Time, Baseline | 110
  Q7: A Little/None of the Time, Week 26 | 228
  Q7: A Little/None of the Time, Week 52 | 226
  Q7: Missing, Baseline | 2
  Q7: Missing, Week 26 | 2
  Q7: Missing, Week 52 | 0

9. Secondary Outcome: Number of Participants With Change in Concomitant Medication of Osteoarthritis Therapy at Week 52
Description: Participants were asked about their perception regarding any additional Osteoarthritis medications or treatments or any changes in regimen or dosages compared to their baseline (Day 0) state. Any change in the therapy (increased therapy, decrease therapy, no change in therapy) during the study was reported.
Time Frame: Baseline up to Week 52
Population: ITT population. Number of participants analysed = participants with baseline and Week 52 data.
Measure: Number; unit: participants
Arm/Group | Synvisc-One
Number analyzed (Participants) | 369
participants
  Increased Therapy | 5
  Decreased Therapy | 2
  No Change in Therapy | 362

10. Secondary Outcome: Time Between Initial and Repeat Synvisc-One Treatment
Description: Time Between initial and repeat Synvisc-One Treatment was duration between initial and repeat injection in those participants who received repeat injection.
Time Frame: Baseline up to Week 52
Population: ITT population. Number of participants analysed = participants from ITT population who received repeat injection.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Synvisc-One
Number analyzed (Participants) | 11
weeks | 38.31 (13.403)

11. Secondary Outcome: Change From Baseline in WOMAC A1 Subscore After Repeat Injection
Description: WOMAC is health status measure questionnaire comprising 3 subscales (pain, stiffness and physical function). WOMAC A1 (measure of pain during walking on a flat surface) was measured using a visual analogue scale (100 mm line marked by participants with total score ranging from 0-100). Lower score represents lower pain. Data are reported for those participants who received repeat injection. Here, baseline represents the day at which a participant received repeat injection (Week 26, 39 or 52).
Time Frame: Baseline; Weeks 1, 4 after repeat injection (missing data imputed by LOCF)
Population: Repeat Intent to treat population included all participants who were eligible for repeat treatment and received at least one repeat dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc-One
Number analyzed (Participants) | 11
units on a scale
  Week 1 After Repeat Injection | -12.4 (15.32)
  Week 4 After Repeat Injection | -10.1 (13.05)

12. Secondary Outcome: Change From Baseline in WOMAC A Score After Repeat Injection
Description: WOMAC is health status measure questionnaire comprising 3 subscales (pain, stiffness and physical function). WOMAC A (measure of pain) calculated as a mean of 5 individual components, measured using a visual analogue scale (100 mm line marked by participants with score ranging from 0-100). Total score range is 0 to 100, where higher scores indicate higher pain. Data are reported for those participants who received repeat injection. Here, baseline represents the day at which a participant received repeat injection (Week 26, 39 or 52).
Time Frame: Baseline; Weeks 1, 4 after repeat injection (missing data imputed by LOCF)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc-One
Number analyzed (Participants) | 11
units on a scale
  Week 1 After Repeat Injection | -4.04 (10.571)
  Week 4 After Repeat Injection | -3.05 (13.473)

13. Secondary Outcome: Change From Baseline in WOMAC B Score After Repeat Injection
Description: WOMAC is health status measure questionnaire comprising 3 subscales (pain, stiffness and physical function). WOMAC B (measure of stiffness) calculated as a mean of 2 individual components, measured using a visual analogue scale (100 mm line marked by participants with score ranging from 0-100). Total score range is 0 to 100, where higher scores indicate higher stiffness. Stiffness is defined as a sensation of decreased ease in movement of joint. Data are reported for those participants who received repeat injection. Here, baseline represents the day at which a participant received repeat injection (Week 26, 39 or 52).
Time Frame: Baseline; Weeks 1, 4 after repeat injection (missing data imputed by LOCF)
Population: Repeat intent to treat population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc-One
Number analyzed (Participants) | 11
units on a scale
  Week 1 After Repeat Injection | -6.14 (6.034)
  Week 4 After Repeat Injection | -3.23 (12.009)

14. Secondary Outcome: Change From Baseline in WOMAC C Score After Repeat Injection
Description: WOMAC is health status measure questionnaire comprising 3 subscales (pain, stiffness and physical function). WOMAC C (measure of physical function) calculated as a mean of 17 individual components, measured using a visual analogue scale (100 mm line marked by participants with score ranging from 0-100). Total score range is 0 to 100, where higher scores indicate higher worse function. Physical function refers to participant's ability to move around and perform usual activities of daily living. Data are reported for those participants who received repeat injection. Here, baseline represents the day at which a participant received repeat injection (Week 26, 39 or 52).
Time Frame: Baseline; Weeks 1, 4 after repeat injection (missing data imputed by LOCF)
Population: Repeat intent to treat population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synvisc-One
Number analyzed (Participants) | 11
units on a scale
  Week 1 After Repeat Injection | -4.08 (7.578)
  Week 4 After Repeat Injection | -4.66 (6.005)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final follow up visit (up to Week 56) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent AEs that is AEs that developed/worsened during the 'on treatment period' (From First dose of study drug until the end of study period). Analysis performed on safety population included all participants treated in the study. Data was planned to be reported for systemic and local adverse events separately.
Groups:
- Synvisc-One: Systemic Adverse Event: Single 6 mL IA injection of Synvisc-One at Day 0 (Initial Treatment). Participants received repeat injection based on physician's discretion of safety and efficacy at Week 26, 39 or 52 (Repeat treatment). Repeat injection was given if there was no major safety concerns and WOMAC A1 subscore (measurement of pain while walking on flat surface) was between 40-80 mm (at Week 26, 39 or 52) when measured on a 0-100 mm scale, where higher score indicate higher pain.Systemic adverse events were defined as any adverse event which occurred anywhere other than in the treated joint.
- Synvisc-One: Local Adverse Event: Single 6 mL IA injection of Synvisc-One at Day 0 (Initial Treatment). Participants received repeat injection based on physician's discretion of safety and efficacy at Week 26, 39 or 52 (Repeat treatment). Repeat injection was given if there was no major safety concerns and WOMAC A1 subscore (measurement of pain while walking on flat surface) was between 40-80 mm (at Week 26, 39 or 52) when measured on a 0-100 mm scale, where higher score indicate higher pain. Local adverse events were defined as any adverse event which occurred in the treated joint.
Arm/Group | Synvisc-One: Systemic Adverse Event | Synvisc-One: Local Adverse Event
Serious Adverse Events (participants affected / at risk) | 5/394 | 1/394
Other Adverse Events (participants affected / at risk) | 23/394 | 22/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synvisc-One: Systemic Adverse Event (N=394) | Synvisc-One: Local Adverse Event (N=394)
Cardiac arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0
Myelomalacia (Nervous system disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synvisc-One: Systemic Adverse Event (N=394) | Synvisc-One: Local Adverse Event (N=394)
Constipation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 4 | 0
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Head discomfort (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.